CLINICAL TRIAL: NCT00184561
Title: Change in HbA1c With Biphasic Insulin Aspart 70/30 in Two Different Treatment Regiments in Subjects With Type 2 Diabetes Inadequately Controlled With Oral Anti-diabetic Drug Therapy.
Brief Title: Effectiveness and Safety of Biphasic Insulin Aspart 70/30 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1707
Record Dates: First submitted 2005-08-29; First posted 2005-09-16 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart

SUMMARY:
This trial is conducted in Asia. This is a clinical trial investigating the effectiveness of using Biphasic Insulin Aspart 70/30 in two different treatment regiments for 6 months in subjects with type 2 diabetes, not well controlled on their current oral anti-diabetic drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1C = 7.5%
* Insulin naïve
* Current treatment by Oral Anti-diabetic Drugs

Exclusion Criteria:

* Severe medical conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2005-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | After 24 weeks of treatment

SECONDARY OUTCOMES:
Adverse events
Weight change
Fasting blood glucose
Hypoglycaemic episodes
2-hour postprandial blood glucose
after 24 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (7):
- China (7):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Wuhan, Hubei
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality

REFERENCES:
- [Result] Yang W, Ji Q, Zhu D, Yang J, Chen L, Liu Z, Yu D, Yan L. Biphasic insulin aspart 30 three times daily is more effective than a twice-daily regimen, without increasing hypoglycemia, in Chinese subjects with type 2 diabetes inadequately controlled on oral antidiabetes drugs. Diabetes Care. 2008 May;31(5):852-6. doi: 10.2337/dc07-1992. Epub 2008 Feb 11. PMID 18268073
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com